CLINICAL TRIAL: NCT03453697
Title: Effects of Acute Intermittent Hypoxia on Brain Function Imaging and Systemic Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XH-17-016
Record Dates: First submitted 2018-02-07; First posted 2018-03-05 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Hypoxemia
Keywords: Intermittent Hypoxemia; diffusion tensor imaging; oxidative stress
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acute intermittent hypoxia (Experimental): Adjust the proportion of nitrogen and oxygen, through increasing the suction nitrogen concentration, the subject's blood oxygen saturation could decrease to 80%~90% within 30 seconds and also lasts 30 seconds; then quickly reduce the concentration of nitrogen gas suction to make the subject's blood oxygen saturation gradually return to normal level (consistent with the air inhalation), and then continue breathing air about 60 seconds to enter the next round of hypoxic state.Through adjusting the inhaled nitrogen concentration in patients, the patients could be simulated as the OSA patients who had intermittent hypoxic state due to upper airway collapse at night. This process is equivalent to acute intermittent hypoxia 25-30 times/h, which is clinically intermediate to severe OSA.
  Interventions: Device: acute intermittent hypoxia

INTERVENTIONS:
Device: acute intermittent hypoxia — Adjust the proportion of nitrogen and oxygen, through increasing the suction nitrogen concentration, the subject's blood oxygen saturation could decrease to 80%~90% within 30 seconds and also lasts 30 seconds; then quickly reduce the concentration of nitrogen gas suction to make the subject's blood oxygen saturation gradually return to normal level (consistent with the air inhalation), and then continue breathing air about 60 seconds to enter the next round of hypoxic state.

SUMMARY:
Effects of acute intermittent hypoxia on brain function imaging and systemic inflammation

Patients with obstructive sleep apnea (OSAS) may have neurological cognitive impairment. The reason is not clear. Intermittent hypoxia is one of the main manifestations of OSAS.

The investigators hypothesize that acute intermittent hypoxia (AIH) can lead to abnormal metabolic activity in some regions of the brain, which may be associated with systemic inflammation.

The investigators proposed in 12 to 15 cases of healthy volunteers, in the form of breathing in the nitrogen intermittently, were observed before and after AIH MRI diffusion tensor imaging (DTI) changes in brain regions and at the same time understand the inflammatory factors and the change of oxidative stress in the human body.

The investigators look at the data from different brain regions of the brain DTI anisotropic score (FA), radial diffusion coefficient (RD), axial diffusion coefficient (AD) and peripheral blood interleukin-6 (IL - 6), interleukin-8 (IL - 8), interleukin-10(IL - 10), tumor necrosis factor alpha (TNF-α), Interleukin-1 beta (IL-1β), Leptin, high sensitivity reactive protein‭‬‬‬‬(hsCRP), Intercellular Adhesion Molecule 1(ICAM 1),Vascular cell adhesion protein 1(VCAM-1) , E-selectin, endothelin-1(ET - 1), 8-iso-PGF2α,3-nitrotyrosine(3-NT),hypoxia-inducible factor 1α(HIF 1α).

Statistical data processing includes: the matching t test of the above indicators before and after AIH; The relationship between DTI and peripheral blood inflammatory factors was analyzed by single factor. Using DTI as the dependent variable, the peripheral blood inflammatory factor was analyzed by multifactor correlation.

Ultimately, the effect of AIH on the brain's regional functions will be understood, and whether the effect is related to systemic inflammation.

DETAILED DESCRIPTION:
In this study, the potential risks to subjects and their corresponding prevention measures:

1. During the test, the volunteers may feel mild sleepiness due to oxygen. (Countermeasures: the subjects have a rest in bed, avoid activity, carry out the whole-process pulse oxygen and heart-rate blood pressure monitoring, and have the full care of the practicing physician)
2. Venous blood is extracted pre- and post-test, and a few subjects may have halo bloody phenomenon. (Countermeasures: inform, select and remove the halo blood volunteers prior to test.)
3. During the test, two MRI scans were performed and each was 20 minutes; the duration was longer than the general MRI (no risk).

Judging criteria for adverse events： According to researchers' own experiment, the low oxygen state had no adverse effects on the body or had only slight fatigue and somnolence, which could be improved after inhaling oxygen.

Plan to recruit and enroll 15 healthy volunteers Group time: March 2018 to March 2019 Follow-up time: the last volunteer was followed up for 1 month after completing the test.

Testing method：

1. Smoking, alcohol drinking, overeating, staying up late were all prohibited one week before the test.
2. The recruiter came to the test center on the testing morning, and the blood was extracted to check the following: blood routine, hsCRP, blood IL-6, IL-8, TNF-α, IL-1β, leptin , ICAM-1, VCAM-1, E-selectin, ET-1, etc.

   The doctor will check volunteers' EKG as well as their blood pressure, heart rate, respiration rate, blood oxygen saturation (when inhaling air). The first DTI was scanned and also process their dataset.
3. Then, the test formally started and immediately entered the intermittent hypoxia cycle: With a mouth-nose mask, which can adjust the proportion of nitrogen and oxygen, the doctor could monitor the blood oxygen saturation; through increasing the suction nitrogen concentration, the subject's blood oxygen saturation could decrease to 80%~90% within 30 seconds and also lasts 30 seconds; then quickly reduce the concentration of nitrogen gas suction to make the subject's blood oxygen saturation gradually return to normal level (consistent with the air inhalation), and then continue breathing air about 60 seconds to enter the next round of hypoxic state.

Through adjusting the inhaled nitrogen concentration in patients, the patients could be simulated as the OSA patients who had intermittent hypoxic state due to upper airway collapse at night. This process is equivalent to AIH 25-30 times/h, which is clinically intermediate to severe OSA.

The subjects always keep quiet and undisturbed during the experiment. The low oxygen cycle totally lasted six hours.

4．Subsequently, the subjects repeated the relevant blood tests (Experiment 2) and related checks, and accepted the second DTI scan for comparison with the first scan.

All blood samples in the test are backup. If the testing results appeared obvious abnormality, they can be reviewed immediately. The MRI examination before and after hypoxia was completed on the same day of the test and immediately uploaded to the imaging system, so there would be no data loss. If the subjects felt uncomfortable during the test, they could quit the test at any time. The investigators will re-recruit new qualified participants to carry out the test.

Statistical data processing includes: (1) the paired t-test with the above indicators pre- and post-AIH; (2) the relationship between DTI measures and peripheral blood inflammatory factors by single factor analysis. (3) Using DTI as the dependent variable and the peripheral blood inflammatory factor as the independent variable, multifactor correlation was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 50 years old, no physical abnormalities
* Without both smoking and drinking habits
* Without the following symptoms: heart, lung, liver, kidney, and thyroid diseases; neuropsychiatric disorders, diabetes history; histories of craniocerebral surgery and tumor disease; recent acute infectious disease (2 weeks); diseases of chronic systemic infection and inflammation
* BMI index in the normal range
* Without snoring and sleep apnea
* No metal in vivo implantation

Exclusion Criteria:

* Diseases such as OSAS or other sleep apnea
* Recent craniocerebral trauma (1 month)
* Alcohol abuse and psychotropic drugs
* EKG checking abnormality or previous history of chest tightness palpitations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Fractional anisotropy | One year
  Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions. FA is a measure often used in diffusion imaging where it is thought to reflect fiber density, axonal diameter, and myelination in white matter. The FA is an extension of the concept of eccentricity of conic sections in 3 dimensions, normalized to the unit range.

CONTACTS AND LOCATIONS:
Overall Officials: Song Liu, M.d., Ph.D., Study Director — Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No